CLINICAL TRIAL: NCT02827656
Title: Luteal Phase Support With Human Chorionic Gonadotropin (hCG) Versus Gonadotropin Releasing Hormone (GnRh) Agonist in IVF Patients Who Are Risk for Developing OHSS
Brief Title: Comapring Luteal Phase Support in IVF Patients Who Are at High Risk for Developing OHSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 056-16MMC
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
Keywords: Fertilization in vitro; Luteal Phase; ovarian hyperstimulation syndrome
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decapeptyl support (Experimental): S.C single luteal Decapeptyl 0.1 mg on days 3, 6,9 post ovulation triggering
  Interventions: Drug: Decapeptyl
- hCG luteal support (Active Comparator): S.C single luteal S.C recombinant hCG 50 micrograms on days 3 ovulation triggering
  Interventions: Drug: hCG luteal support

INTERVENTIONS:
Drug: Decapeptyl — luteal support as described and vaginal progesterone 200 mg 3 times a day
  Arms: Decapeptyl support
Drug: hCG luteal support — luteal support as described and vaginal progesterone 200 mg 3 times a day
  Arms: hCG luteal support

SUMMARY:
The purpose of this study is to compare two luteal support protocols in In vitro fertilization patients (IVF) and are at risk of developing ovarian hyperstimulation syndrome (OHSS). We would like to determine whether luteal Decapeptyl on days 3, 6,9 post ovulation triggering is as good as low dose hCG on day 3 post triggering..

DETAILED DESCRIPTION:
This is randomized clinical trial studying two luteal support protocols of In vitro fertilization patients (IVF) treated by a GnRH antagonist (GnRH ant) protocol and are at risk of developing ovarian hyperstimulation syndrome (OHSS). The randomization procedure will be performed by a third party in the hospital by using a randomization table: patients fulfilling the inclusion and exclusion criteria and giving their informed consent will be randomized into one of two arms. This study does not include any intervention affecting the ovarian stimulation and is solely intended to test the post ova pickup period.

One arm will be treated by luteal Decapeptyl on days 3, 6,9 post ovulation triggering. Second arm will be treated by low dose hCG on day 3 post triggering. All patients to be recruited are treated for acceptable IVF indications in Meir medical center (MMC) and their registry is computerized in the general system of MMC. For the purpose of the study we will use the only the data of patients recruited to the study and were giving their informed consent. Each patient recruited will have a unique study identity (ID) . The patients' information will be pooled from the computerized file into an Excel spread sheet: in this Excel file the names will be erased and only the unique study ID will appear. The information regarding the coding key will be kept as a hard copy in a locked room inside the IVF unit in a special study folder. The study was approved by MMC institutional Helsinki board.

The data retrieved for each patients is not unique for the study but includes the basic variables monitored in every IVF cycle : Estradiol serum levels (E2), Progesterone serum levels (P), number of follicles as counted by trans-vaginal ultrasound, endometrial thickness as measured by trans-vaginal ultrasound, Follicle stimulating hormone (FSH) dosing, number of stimulation days, number of eggs retrieved, fertilization rate, blastulation rate, number of embryos transferred, embryo quality, positive pregnancy test, implantation rate, presence of a clinical pregnancy, presence of OHSS. Since these are mandatory variables in the treatment we do not expect any missing data. In addition to these mandatory data the study patients will be performing two additional blood tests on day 3 post ovum pickup and on the transfer day itself (day 5 post ovum pickup) including Estradiol serum levels (E2) and Progesterone serum levels (P).

Outcome measures: Day of transfer Progesterone serum levels, OHSS rate, implantation rate, clinical pregnancy rate.

Sample size calculation based on Kol S et al 2015, regarding the day of transfer Progesterone level (pooled standard deviation: 40nmol/L), alpha of 5%, 80% power, then a non-inferiority study will require 22 patients in each group and a total of 44 patients. Once including an expected 10% chance of freeze all in this population we will include 50 patients.

Statistical analysis: Analysis of data was performed using the SPSS 23.0 computer package (SPSS Inc., Chicago, IL). Normally distributed data were analyzed by student t test . χ2 or Fisher's exact test will be used for comparisons of rates and proportions. All P values were tested as two-sided and considered significant at less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* IVF treatment
* GnRH antagonist protocol
* GnRH agonist triggering of ovulation
* High risk for OHSS as expressed by either E2 serum level >2500 pg/ml

Exclusion Criteria:

* background maternal morbidity
* Any protocol other than GnRH antagonist protocol
* hCG triggering of ovulation
* E2 serum level >4500 pg/ml
* Aspiration of >25 ova
* Embryo transfer prior to day 5

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progesterone serum level | day 5 post ovum pickup

SECONDARY OUTCOMES:
positive pregnancy test | 9-12 days post embryo transfer
implantation rate | 30-33 days post embryo transfer
clinical pregnancy rate | 30-33 days post embryo transfer
  clinical pregnancy is considered as a presence of a viable embryo (heart activity present)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Wiser, MD, Principal Investigator — MMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- [Background] Whelan JG 3rd, Vlahos NF. The ovarian hyperstimulation syndrome. Fertil Steril. 2000 May;73(5):883-96. doi: 10.1016/s0015-0282(00)00491-x. PMID 10785212
- [Background] Humaidan P, Bredkjaer HE, Bungum L, Bungum M, Grondahl ML, Westergaard L, Andersen CY. GnRH agonist (buserelin) or hCG for ovulation induction in GnRH antagonist IVF/ICSI cycles: a prospective randomized study. Hum Reprod. 2005 May;20(5):1213-20. doi: 10.1093/humrep/deh765. Epub 2005 Mar 10. PMID 15760966
- [Background] Griesinger G, Schultz L, Bauer T, Broessner A, Frambach T, Kissler S. Ovarian hyperstimulation syndrome prevention by gonadotropin-releasing hormone agonist triggering of final oocyte maturation in a gonadotropin-releasing hormone antagonist protocol in combination with a "freeze-all" strategy: a prospective multicentric study. Fertil Steril. 2011 May;95(6):2029-33, 2033.e1. doi: 10.1016/j.fertnstert.2011.01.163. Epub 2011 Mar 2. PMID 21371705
- [Background] Kol S, Breyzman T, Segal L, Humaidan P. 'Luteal coasting' after GnRH agonist trigger - individualized, HCG-based, progesterone-free luteal support in 'high responders': a case series. Reprod Biomed Online. 2015 Dec;31(6):747-51. doi: 10.1016/j.rbmo.2015.09.001. Epub 2015 Sep 9. PMID 26507279